CLINICAL TRIAL: NCT07069244
Title: Blood Markers in Periodontal Inflammation and Alzheimer's Disease: A Retrospective Case-Control Study
Brief Title: Investigation of the Relationship Between Periodontitis and Alzheimer's Disease in Terms of Blood Parameters
Status: Completed | Type: Observational
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Kubra Karaduran, Assistant professor, Uskudar University
Other Study IDs: KKARADURAN
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Periodontal Disease; Periodontitis; Periodontal Inflammation; Biomarkers / Blood; Blood Cell Count; Alzheimer Disease
Keywords: Alzheimer disease; biomarkers; blood cell count; complete blood count; periodontal disease; periodontitis
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Periodontitis with Alzheimer's disease
  Interventions: Diagnostic Test: Complete Blood Count Test; Diagnostic Test: Periodontal examinations; Diagnostic Test: Clinical Dementia Rating scale; Diagnostic Test: Standardized Mini-Mental Test
- Control group: Periodontitis without Alzheimer's disease
  Interventions: Diagnostic Test: Complete Blood Count Test; Diagnostic Test: Periodontal examinations

INTERVENTIONS:
Diagnostic Test: Complete Blood Count Test — Complete blood count test provides data on total white blood cell count, neutrophil count, neutrophil percentage, lymphocyte count, lymphocyte percentage, monocyte count, monocyte percentage, eosinophil count, eosinophil percentage, basophil count, basophil percentage, platelet count, platelet distribution width (PDW), mean platelet volume (MPV), plateletcrit (PCT), erythrocyte count, hemoglobin, hematocrit (HCT), mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC) and red blood cell distribution width (RDW). In addition, neutrophil-lymphocyte ratio (NLR), monocyte-lymphocyte ratio (MLR), platelet-leukocyte ratio (PLR), Pan-Immune-Inflammation Value (PIV), Systemic Immune-Inflammation Index (SII), Hemoglobin-to-Red Cell Distribution Width Ratio (HRR) values are also formulated from these parameters.
Diagnostic Test: Periodontal examinations — With periodontal evaluation, plaque percentage, probing pocket depth, percentage of bleeding on probing, clinical attachment level, number of teeth, periodontal inflammatory surface area (PISA) parameters are recorded.
Diagnostic Test: Clinical Dementia Rating scale — Stage I: mild Alzheimer's disease, Stage II: moderate Alzheimer's disease, Stage III: severe Alzheimer's disease
  Groups: Case group
Diagnostic Test: Standardized Mini-Mental Test — Cognitive status is assessed with the Standardized Mini-Mental Test.
  Groups: Case group

SUMMARY:
The aim of this study was to analyse the possible relationship between periodontal inflammation and Alzheimer's disease and to investigate the role of blood parameters in this relationship.

DETAILED DESCRIPTION:
This retrospective case-control study will include individuals who were clinically and radiographically examined, diagnosed with periodontal disease, read and signed informed consent forms between March 2022 and July 2025 at the Periodontology Departments of Bezmialem Vakif University, Uskudar University and Bolu Abant Izzet Baysal University Faculty of Dentistry.

In this study, two groups will be formed as a case group consisting of individuals with periodontitis diagnosed with probable Alzheimer's disease according to NINCDS-ADRDA and DSM-V diagnostic criteria and a control group consisting of individuals with periodontitis only.

Patients who underwent periodontal evaluations at six sites per tooth, with the following parameters recorded-plaque percentage, probing pocket depth, percentage of bleeding on probing, clinical attachment level, number of teeth, and periodontal inflamed surface area (PISA)-will be included in the study.

Compliance with the inclusion and exclusion criteria will be verified through patient files and digital records. In individuals with a probable diagnosis of Alzheimer's disease according to NINCDS-ADRDA and DSM-V diagnostic criteria, disease stage as determined by the Clinical Dementia Rating scale and Standardized Mini-Mental Test (SMMT) scores will also be recorded.

Hematological data will be obtained from patients' recorded complete blood count test results and the following parameters will be utilized:

* White blood cell count, neutrophil, lymphocyte, monocyte, eosinophil, basophil counts and percentages, neutrophil/lymphocyte ratio (NLR), monocyte/lymphocyte ratio (MLR)
* Platelet count, platelet/lymphocyte ratio (PLR), platelet distribution width (PDW), mean platelet volume (MPV), plateletcrit (PCT)
* Erythrocyte count, hemoglobin (HGB), hematocrit (HCT), mean corpuscular volume (MCV), mean corpuscular haemoglobin (MCH), mean corpuscular haemoglobin concentration (MCHC), red blood cell distribution width (RDW)
* In addition, inflammation indicators such as pan-immune inflammation value (PIV), systemic immune-inflammation index (SII) and hemoglobin/erythrocyte ratio (HRR), which are formulated from the above parameters, will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Between March 2022 and July 2025, those who applied to the Periodontics Departments of the Dentistry Faculties of Uskudar University, Bezmialem Vakif University and Bolu Abant Izzet Baysal University,
* Informed consent form was obtained during the examination,
* Over 50 years of age,
* Non-smoker and non-alcoholic,
* No psychiatric disorders affecting cognitive status and no medication affecting cognitive status,
* Complete blood count was performed within the 6 months prior to the date of inclusion in the study,
* No dental treatment within the last 1 year,
* Periodontal examination was performed by expert periodontologists who calibrated the inter- and intra-examination,
* Individuals diagnosed with periodontitis as a result of periodontal examination and radiographic examination, and
* For individuals diagnosed with Alzheimer's disease: Recording their stage according to the Clinical Dementia Rating (CDR) and Standardized Mini-Mental Test (SMMT) scores

Exclusion Criteria:

* Individuals with fewer than 10 teeth,
* Individuals with uncontrolled systemic disease,
* Individuals who regularly use anti-inflammatories or corticosteroids

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with periodontitis with Alzheimer's disease (Case group), Individuals with periodontitis without Alzheimer's disease (Control group)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-08-05 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Probing pocket depth | Baseline
  Measurement of the depth of a sulcus or periodontal pocket determined by measuring distance from a gingival margin to the base of the sulcus or pocket with a calibrated periodontal probe.
Bleeding on probing (BOP) | Baseline
  The number obtained by dividing the sum of the positive areas by the sum of the examined areas is multiplied by 100 and the value obtained is expressed as the percentage of bleeding at probing (BOP%).
Periodontal inflammatory surface area (PISA) | Baseline
  It is the calculation of the area of ulcerated periodontal pockets showing bleeding on probing based on the periodontal epithelial surface area.

SECONDARY OUTCOMES:
Clinical attachment level | Baseline
  Clinical attachment level (CAL) is a more reliable indicator of periodontal support around a tooth than probing depth alone, as it is measured from a fixed anatomical landmark-the cementoenamel junction (CEJ)-which remains constant over time.
  Calculating CAL requires two measurements: the distance from the gingival margin to the CEJ and the probing depth.
  In cases of gingival recession, CAL is calculated by adding the probing depth to the distance from the gingival margin to the CEJ.
  In cases of gingival overgrowth, CAL is determined by subtracting the distance from the gingival margin to the CEJ from the probing depth.
Plaque percentage | Baseline
  The presence or absence of plaque is determinant, recorded as (+) in the presence of plaque or (-) in the absence of plaque, and the percentage of the entire mouth affected by plaque is expressed as a percentage (P%).
Number of teeth | Baseline
  Recording the number of teeth present
White blood cell count | Between baseline and -6th month
  White blood cell (WBC) count measures the total number of leukocytes in peripheral blood, usually expressed as cells per microliter (cells/µL). WBC is essential for evaluating immune status, infections, and inflammatory conditions.
Neutrophil count | Between baseline and -6th month
  Neutrophil count measures the absolute number of neutrophils in peripheral blood, typically expressed as cells per microliter (cells/µL). Neutrophils play a critical role in innate immune defense, especially against bacterial infections.
Lymphocyte count | Between baseline and -6th month
  Lymphocyte count measures the absolute number of lymphocytes in peripheral blood, typically expressed as cells per microliter (cells/µL). Lymphocytes are essential for adaptive immune responses and immune memory.
Monocyte count | Between baseline and -6th month
  Monocyte count measures the absolute number of monocytes in peripheral blood, typically expressed as cells per microliter (cells/µL). Monocytes are key cells in immune response, inflammation, and tissue repair.
Eosinophil count | Between baseline and -6th month
  Eosinophil count measures the absolute number of eosinophils in peripheral blood, typically expressed as cells per microliter (cells/µL). Eosinophils are involved in allergic responses and parasitic infections.
Basophil count | Between baseline and -6th month
  Basophil count measures the absolute number of basophils in peripheral blood, usually expressed as cells per microliter (cells/µL). Basophils are involved in allergic and inflammatory responses.
Percentage of neutrophils | Between baseline and -6th month
  The percentage of neutrophils represents the proportion of neutrophils among total white blood cells, expressed as a percentage (%). Neutrophils are key players in innate immune response and bacterial defense.
Percentage of lymphocytes | Between baseline and -6th month
  The percentage of lymphocytes indicates the proportion of lymphocytes among total white blood cells, expressed as a percentage (%). Lymphocytes are essential for adaptive immune responses.
Percentage of monocytes | Between baseline and -6th month
  The percentage of monocytes represents the proportion of monocytes among total white blood cells, expressed as a percentage (%). Monocytes play a critical role in immune response, inflammation, and tissue repair.
Percentage of eosinophils | Between baseline and -6th month
  The percentage of eosinophils indicates the proportion of eosinophils among total white blood cells, expressed as a percentage (%). Eosinophils play key roles in allergic responses and parasitic infections.
Percentage of basophils | Between baseline and -6th month
  The percentage of basophils represents the proportion of basophils among total white blood cells, usually expressed as a percentage (%). Basophils are involved in allergic and inflammatory responses.
Platelet count (PLT) | Between baseline and -6th month
  Platelet count (PLT) measures the number of platelets in a given volume of blood, expressed in thousands per microliter (×10³/μL). It is essential for assessing clotting function, bleeding disorders, and inflammatory status.
Platelet distribution width (PDW) | Between baseline and -6th month
  Platelet Distribution Width (PDW) measures the variability in platelet size, reflecting platelet heterogeneity. It is used to assess platelet activation, production disorders, and systemic inflammatory conditions.
Mean platelet volume (MPV) | Between baseline and -6th month
  Mean Platelet Volume (MPV) measures the average size of platelets in the blood and is expressed in femtoliters (fL). It reflects platelet activation and production and is used to assess platelet-related disorders and systemic inflammation.
Plateletcrit (PCT) | Between baseline and -6th month
  Plateletcrit (PCT) represents the volume percentage of platelets in the blood and is calculated by multiplying the platelet count by the mean platelet volume. It reflects platelet mass and is used to assess platelet-related disorders and systemic inflammatory status.
Red blood cell count | Between baseline and -6th month
  Red blood cell (RBC) count measures the number of erythrocytes in a given volume of blood, typically expressed in million cells per microliter (×10⁶/μL). It is used to assess oxygen transport capacity, anemia, and overall hematologic health.
Hemoglobin (Hb) | Between baseline and -6th month
  Hemoglobin is the iron-containing protein in red blood cells responsible for transporting oxygen throughout the body. Hemoglobin concentration is measured in g/dL and is commonly used to assess anemia and systemic health status.
Hematocrit (HCT) | Between baseline and -6th month
  Hematocrit (HCT) represents the percentage of whole blood volume occupied by red blood cells. It is used to evaluate oxygen-carrying capacity, anemia status, and hydration level.
Mean corpuscular volume (MCV) | Between baseline and -6th month
  Mean Corpuscular Volume (MCV) indicates the average size of red blood cells and is expressed in femtoliters (fL). It is used to classify types of anemia.
Mean corpuscular hemoglobin (MCH) | Between baseline and -6th month
  Mean Corpuscular Hemoglobin (MCH) represents the average amount of hemoglobin per red blood cell. It is commonly used to classify types of anemia.
Mean corpuscular hemoglobin concentration (MCHC) | Between baseline and -6th month
  Mean Corpuscular Hemoglobin Concentration (MCHC) reflects the average concentration of hemoglobin in red blood cells and is expressed in g/dL. It is used to assess anemia types.
Red blood cell distribution width (RDW) | Between baseline and -6th month
  Red Cell Distribution Width (RDW) reflects the variability in size of circulating red blood cells. It is considered a potential marker of inflammation, oxidative stress, and chronic disease burden.
Neutrophil-to-lymphocyte ratio (NLR) | Between baseline and -6th month
  The neutrophil-to-lymphocyte ratio (NLR) is calculated by dividing the absolute neutrophil count by the absolute lymphocyte count. It serves as a marker of systemic inflammation and immune system balance
Monocyte-to-Lymphocyte Ratio (MLR) | Between baseline and -6th month
  Monocyte-to-Lymphocyte Ratio (MLR) is the ratio of monocyte count to lymphocyte count in peripheral blood. It is used as a marker of systemic inflammation and immune system balance in various diseases.
Platelet-to-lymphocyte ratio (PLR) | Between baseline and -6th month
  The platelet-to-lymphocyte ratio (PLR) is a systemic inflammation marker calculated by dividing the absolute platelet count by the absolute lymphocyte count.
Pan-immune inflammation value (PIV) | Between baseline and -6th month
  It is a biomarker that evaluates the immune system and inflammation together. PIV= (Neutrophils × Monocytes × Platelets) / Lymphocytes
Systemic immune-inflammation index (SII) | Between baseline and -6th month
  It is a parameter reflecting systemic inflammation and immune response. SII= (Neutrophil × Platelet) / Lymphocyte
Hemoglobin to erythrocyte ratio (HRR) | Between baseline and -6th month
  It shows the ratio between the haemoglobin level and the distribution width of red blood cells.
  HRR= Hemoglobin / RDW
Standardized Mini-Mental Test (SMMT) | Baseline
  The SMMT is used to quantitatively assess cognitive status in Alzheimer's disease patients. The maximum score of the SMMT is 30, of which 10 points correspond to orientation questions, 3 points to recording memory, 5 points to attention and calculation, 3 points to recall and 9 points to language.
Clinical Dementia Rating Scale | Baseline
  The Clinical Dementia Rating (CDR) Scale is used to stage different types of dementia, especially Alzheimer-type dementia.
  Stage I: Mild, Satege II: Moderate, Stage III: Severe

CONTACTS AND LOCATIONS:
Overall Officials: OZLEM GELISIN, Study Chair — Dr. Sadi Konuk Training and Research Hospital; AHMET AYDOGDU, Study Chair — Istanbul Galata University; SADIYE GUNPINAR, Study Chair — Bezmialem Vakif University; ZEYNEP AKGUL, Study Chair — Abant Izzet Baysal University; KUBRA KARADURAN, Principal Investigator — Uskudar University
Locations (3):
- Turkey (Türkiye) (3):
  - Bolu Abant Izzet Baysal University, Bolu
  - Bezmialem Vakif University, Istanbul
  - Uskudar University, Istanbul

REFERENCES:
- [Background] Wang RH, Wen WX, Jiang ZP, Du ZP, Ma ZH, Lu AL, Li HP, Yuan F, Wu SB, Guo JW, Cai YF, Huang Y, Wang LX, Lu HJ. The clinical value of neutrophil-to-lymphocyte ratio (NLR), systemic immune-inflammation index (SII), platelet-to-lymphocyte ratio (PLR) and systemic inflammation response index (SIRI) for predicting the occurrence and severity of pneumonia in patients with intracerebral hemorrhage. Front Immunol. 2023 Feb 13;14:1115031. doi: 10.3389/fimmu.2023.1115031. eCollection 2023. PMID 36860868
- [Background] An P, Zhou X, Du Y, Zhao J, Song A, Liu H, Ma F, Huang G. Association of Neutrophil-Lymphocyte Ratio with Mild Cognitive Impairment in Elderly Chinese Adults: A Case-control Study. Curr Alzheimer Res. 2019;16(14):1309-1315. doi: 10.2174/1567205017666200103110521. PMID 31902361
- [Background] Zhou C, Liu Y, Bai J, Luo Y, Song J, Feng P. Mean platelet volume is associated with periodontitis: a cross-sectional study. BMC Oral Health. 2024 Apr 16;24(1):461. doi: 10.1186/s12903-024-04223-8. PMID 38627719
- [Background] Leira Y, Carballo A, Orlandi M, Aldrey JM, Pias-Peleteiro JM, Moreno F, Vazquez-Vazquez L, Campos F, D'Aiuto F, Castillo J, Sobrino T, Blanco J. Periodontitis and systemic markers of neurodegeneration: A case-control study. J Clin Periodontol. 2020 May;47(5):561-571. doi: 10.1111/jcpe.13267. Epub 2020 Mar 12. PMID 32027386
- [Background] Tosatti JAG, Pereira JD, Loures CMG, Fraga VG, Magalhaes CA, Eugenio RDAC, Guimaraes HC, Resende EPF, de Souza LC, Carvalho MDG, Caramelli P, Gomes KB. Complete blood count and systemic inflammation indices in individuals with Alzheimer's disease: A case-control study. J Clin Neurosci. 2025 Feb;132:111011. doi: 10.1016/j.jocn.2024.111011. Epub 2024 Dec 28. PMID 39733506